CLINICAL TRIAL: NCT01057303
Title: EVI-1 Expression in Pediatric AML With 11q23 Abnormalities
Brief Title: Studying Gene Expression in Tissue Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B15; COG-AAML10B15 (Other: Children's Oncology Group); CDR0000664144 (Other: Clinical Trials.gov); NCI-2011-02205 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at gene expression in tissue samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine mRNA from pediatric patients with acute myeloid leukemia with 11q23 translocations by reverse transcriptase-PCR to quantify expression of EVI1 splice variants.

OUTLINE: Cryopreserved mRNA from diagnostic samples is analyzed for gene expression by reverse transcriptase-PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pediatric acute myeloid leukemia with 11q23 abnormalities

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of pediatric acute myeloid leukemia with 11q23 abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Quantification of the expression of EVI1 splice variants

CONTACTS AND LOCATIONS:
Overall Officials: Amy Heerema-McKenney, MD, Principal Investigator — Stanford University